CLINICAL TRIAL: NCT01115205
Title: Assessment of Feasibility and Efficacy of a Project Aimed to Improve Metabolic Control in Type 2 Diabetes Through Lifestyle Changes and Self-monitoring of Blood Glucose
Brief Title: Supervised Walking Groups as a Model to Increase Physical Activity in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Paolo Moghetti, Department of Medicine, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 1264
Record Dates: First submitted 2010-04-26; First posted 2010-05-04 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes
Keywords: Exercise, Walking, Type 2 diabetes, Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised walking groups (Experimental): Patients included in walking groups, under the supervision of a qualified personal trainer.
  Interventions: Behavioral: Supervised walking
- Controls (Active Comparator): Patients receiving the standard counselling procedures of the Verona Diabetic Clinic.
  Interventions: Behavioral: Standard counselling procedure

INTERVENTIONS:
Behavioral: Supervised walking — Walk training, 3 sessions per week for 4 months, under the supervision of a qualified personal trainer.
  Arms: Supervised walking groups
Behavioral: Standard counselling procedure — Verbal and written information about the benefits of exercise and instructions aimed to encourage physical activity. In addition, one group session of counselling on these issues.
  Arms: Controls

SUMMARY:
The purpose of the study is to evaluate the impact of an exercise programme organized into supervised walking groups on metabolic control, functional capacity and overall quantity of physical activity in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Regular, moderate-intensity physical activity can attenuate hyperglycemia in subjects with type 2 diabetes. In addition, these programmes may favourably affect several other cardiovascular risk factors in these subjects. However, it still remains unclear how this evidence can be transferred into clinical practice, considering the very large number of diabetic patients and the characteristics of this population, made up predominantly of elderly, sedentary and overweight patients. In this regard, a realistic approach to this issue requires simple and easily available intervention models.

Walking is a typical mild-moderate aerobic physical activity which is easy to organize and does not require specific skills or preliminary sophisticated medical evaluations. This activity could therefore fit well with the need of involvement of large numbers of patients in different logistic situations. However, it has been reported that, due to the low walking speed typical of type 2 diabetic subjects, self-paced walking is inadequate to obtain a significant metabolic improvement in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* diabetes known for at least 2 yr
* physical inactivity
* haemoglobin (Hb)A1c between 6.5-9.9%
* treatment with oral hypoglycaemic agents alone or associated with a bed-time insulin injection
* willingness to participate in a programme of regular physical activity

Exclusion Criteria:

* moderate-severe autonomic or somatic neuropathy
* severe lower limb vasculopathy
* pre-proliferative or proliferative active retinopathy
* moderate to severe chronic renal failure
* unstable angina or recent (in the previous 3 months) myocardial infarction
* acute intercurrent diseases
* acute metabolic decompensation (blood glucose >300 mg/dl or ketonuria in two consecutive checks)
* use of beta-blocker drugs
* subjects unable to complete a 6-min walk test

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in haemoglobin A1c (HbA1c) levels | 4 months
  The measurement of HbA1c is carried out with a DCCT-aligned method.

SECONDARY OUTCOMES:
Change in Body weight | 4 months
Change in Fasting plasma glucose levels | 4 months
Change in Total Cholesterol levels | 4 months
Change in HDL Cholesterol levels | 4 months
Change in LDL Cholesterol levels | 4 months
Change in Triglycerides levels | 4 months
Change in Blood Pressure | 4 months
Change in 6 minutes walk distance | 4 months
  This test measures the number of meters that can be walked in 6 minutes over a 30 m course. It is a simple field test to assess aerobic functional capacity.
Change in C-reactive protein levels | 4 months
Change in Energy expenditure through voluntary physical activity | 4 months
  Energy expenditure is estimated through 7-day activity diaries. The intensity of each activity (defined in metabolic equivalents, MET) is multiplied by duration and the product for each activity is summed to give a total activity score in MET hours/week.
Change in Antidiabetic medications | 4 months
  Class and dosage of blood-glucose lowering drugs are recorded before and at the end of the protocol, to assess changes in hypoglycemic medication during the trial.
Compliance with walking sessions | 4 months
  Attendance at the scheduled walking sessions is recorded for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Moghetti, M.D., Ph.D., Principal Investigator — Universita di Verona

REFERENCES:
- [Derived] Negri C, Bacchi E, Morgante S, Soave D, Marques A, Menghini E, Muggeo M, Bonora E, Moghetti P. Supervised walking groups to increase physical activity in type 2 diabetic patients. Diabetes Care. 2010 Nov;33(11):2333-5. doi: 10.2337/dc10-0877. PMID 20980426